CLINICAL TRIAL: NCT04573231
Title: Evaluation of Prostate Specific Membrane Antigen (PSMA) in HER2-negative, Androgen Receptor (AR)-Positive Metastatic Breast Cancer With 18F-DCFPyL PSMA-based PET/CT
Brief Title: Evaluation of PSMA in HER2- AR+ Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0949; A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); Protocol Version 12/12/2025 (Other: UW Madison); NCI-2020-07434 (Registry Identifier: NCI CTRP); 2020-0949 (Other: UW Madison)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Intervention Model Description: Phase 2, single-center, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL PSMA-based PET/CT (Experimental): * 18F-DCFPyL whole body PET/CT scan
  * Review of relevant imaging and medical record information
  * Blood draw for circulating tumor cells (CTCs)
  * Analysis of diagnostic tissue specimens
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — PSMA is highly expressed on prostate cancer and is associated with metastasis and resistance to anti-androgen therapies. Researchers have evaluated the expression of PSMA in the tumor and tumor-associated neovasculature in primary tumors and distant metastases in patients with breast cancer.

SUMMARY:
The purpose of this research is to determine the expression of prostate specific membrane antigen (PSMA) in human epidermal growth factor receptor 2 (HER2)-negative, androgen receptor (AR)-positive metastatic breast cancer, and to determine its role in resistance to the anti-androgen, bicalutamide. The investigators hypothesize that PSMA expression will correlate with resistance to anti-androgen therapies, as has been documented in prostate cancer, and this can be used to select patients most likely to benefit from these therapies in future clinical trials. 15 people with HER2-negative, AR-positive metastatic breast cancer will be enrolled and be on study for about 3 days.

DETAILED DESCRIPTION:
Primary Objective:

* To evaluate the expression of PSMA via 18F-DCFPyL PSMA-based PET/CT in patients with metastatic HER2-negative, AR-positive breast cancer. Expression of PSMA will be quantified using PSMA-based PET imaging using a novel agent, 18F-DCFPyL, as a non-invasive imaging biomarker of tumor neovasculature in HER2-negative, AR-positive metastatic breast cancer.

Secondary Objectives:

* PSMA PET will be compared with the expression of PSMA in CTCs and diagnostic metastatic tissue from patients with HER2-negative, AR-positive metastatic breast cancer.
* PSMA expression will be correlated with clinical benefit (objective response and progression-free survival) to bicalutamide and ribociclib for patients enrolled in NCT03090165.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with metastatic HER2-negative breast cancer AR expression of ≥ 10%

Exclusion Criteria:

* Other (non-breast) known active malignancy. Participants with previously treated cancers which are in remission or have no evidence of disease are eligible.
* Unable to lie flat during or tolerate PET/CT
* Participants with any medical condition or other circumstances that, in the opinion of the investigator, compromise the safety or compliance of the subject to produce reliable data or completing the study
* Women of childbearing potential must not be pregnant or breast feeding (pregnancy test negative within 7 days prior to PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PSMA Expression as measured by 18F-DCFPyL SUV | up to 3 days
  Quantitative analysis of 18F-DCFPyL PSMA PET uptake will be performed at the lesion-level. Standardized uptake values (SUV) will be measured by manually drawing a region of interest (ROI) to encompass the entire lesion guided by the lesion extent visualized on conventional imaging. PET SUV based quantitative tumor uptake parameters will be obtained.

SECONDARY OUTCOMES:
Expression of PSMA in CTCs | up to 2 weeks
  Expression of PSMA in CTCs will be measured via immunofluorescence.
Expression of PSMA in diagnostic metastatic tissue | up to 3 days
  PSMA expression in tumors will be semi-quantitatively scored by a study pathologist using published methods including separate assessment of tumor-associated and non-tumor vasculature, with the endothelium highlighted by a CD31 immunostain to facilitate definitive recognition.
Change in PSMA Expression on CTCs after 2 weeks of bicalutamide | baseline and up to 2 weeks
  The change in PSMA expression on CTCs will be measured pre and post treatment via immunofluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Fowler, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No